CLINICAL TRIAL: NCT04803565
Title: The Effect of Personalized Shoe Insole on the Gait of Parkinson's Disease Subjects: A Triple-blind Randomized Controlled Trial
Brief Title: The Effect of Personalized Shoe Insole on the Gait of Parkinson's Disease Subjects
Acronym: InsolePD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: JP-002
Record Dates: First submitted 2021-03-04; First posted 2021-03-17 (Actual); Last update posted 2023-10-03 (Actual); Status verified 2023-09

CONDITIONS: Parkinson Disease
Keywords: Parkinson Disease; Foot Orthoses; Randomized controlled trial
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Custom-Made Insole (Experimental): This Group will receive a custom-made shoe insole designed on the foot shape of the subjects.
  The group will also receive Physiotherapy and Occupational Therapy according to current guidelines
  Interventions: Device: Custom-made shoe insole
- Sham Insole (Sham Comparator): This group will receive a Sham shoe insole without any specific custom-made design.
  The group will also receive Physiotherapy and Occupational Therapy according to current guidelines
  Interventions: Device: Sham conventional Insole

INTERVENTIONS:
Device: Custom-made shoe insole — Subjects will receive a custom-made shoe insole designed on the patient's foot and shoes. The subjects should wear the insole for at least 6 hours per day.
  Arms: Custom-Made Insole
Device: Sham conventional Insole — Subjects will receive a conventional insole without any specific property (sham insole)
  Arms: Sham Insole

SUMMARY:
This study aims to assess the efficacy of custom-made shoe insoles, for subjects with Parkinson's Disease (PD).

To do that, a sample of PD subjects has been randomly assigned to an intervention group that will receive the custom-made insoles or a control group that will receive a sham insole without any specific manufacturing.

Both groups will receive Physiotherapy and Occupational Therapy according to PD rehabilitation guidelines.

The principal outcome will be the Time Up&Go test time, secondary outcomes 10 Meters Walking test speed, Berg Balance Scale score, SF12 score, and orthesis liking.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with Idiopathic Parkinson's Disease;
* Age > 18 years;
* Subjects should be in a positive therapeutic window or in the ON phase during the evaluations;
* Subjects must be able to walk at least 10 meters independently with or without any walking aid.

Exclusion Criteria:

* Not clinical stable subjects;
* SUbjects in OFF phase during the evaluations;
* Other neurological conditions (e.g. stroke, peripheral neuropathies, etc.);
* Other pathologies that can negatively influence the subject's walking ability (e.g. surgery at the lower limbs in the previous 6 months, important deformities at the lower limbs, etc.)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2021-03-04 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Change in Time Up&Go test | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Time Up&Go at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))

SECONDARY OUTCOMES:
Change in 10 Meters walking test Speed | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) 10 Meters walking test speed at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Berg Balance Scale Score | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Berg Balance Scale score at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Short-Form12 score | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline Short-form 12 at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Likert scale 4 points | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline Short-form 12 at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test cadence | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test step length | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test step duration | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test stance phase | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test swing phase | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test single support phase | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in 10 Meters Walking Test double support phase | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Kinematic parameters of gait during 10 Meters Walking test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Time Up&Go test sit-to-stand time | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Temporal and kinematic parameters of Time Up&Go test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Time Up&Go test stand-to-sit time | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Temporal and kinematic parameters of Time Up&Go test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Time Up&Go test mid-turning time | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Temporal and kinematic parameters of Time Up&Go test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))
Change in Time Up&Go test end-turning time | Baseline, at 10 weeks, and at 16 weeks.
  Change from Baseline (without insoles (T0) and with insoles (T1)) Temporal and kinematic parameters of Time Up&Go test at 10 weeks (end of outpatient rehabilitation (T2)) and 16 weeks (follow-up (T3))

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Fondazione Don Carlo Gnocchi, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided